CLINICAL TRIAL: NCT02063373
Title: Gait, Stair Climbing and Postural Stability in Knee Osteoarthritis Patients After Hyaluronic Acid Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, nafiseh khalaj, Mrs, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UM/MOHE/HIR D000010-16001
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Bilateral Knee Osteoarthritis
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biomechanis knee OA and HA injection (Experimental): Weekly intra- articular Hyaluronic acid injection (20 MG/ 2 ML) into both knees for five weeks
  Interventions: Other: Hyaluronic acid

INTERVENTIONS:
Other: Hyaluronic acid — treatment: Weekly intra-articular hyaluronic acid injection (20 MG / 2ML) into both knees for five weeks.
  Other Names: Hyalgan; Manufacturer: Fidia Pharmaceutici S.p.A, Italy

SUMMARY:
Treatment: five intro-articular Hyaluronic Acid injection

Assessment has two parts, that are as follow:

1. Postural stability and risk of fall assessment using Biodex stability index and "Timed up and Go" test
2. Gait and stair climbing assessment using Vicon motion capture system synchronized with four force plates.

For knee OA subjects, assessment was done in week one or before injection; and for healthy controls one assessment was performed.

DETAILED DESCRIPTION:
This study aimed to assess the effect of hyaluronic acid injection on Postural stability, biomechanics of gait and stair climbing in individuals with bilateral knee osteoarthritis (OA).

Participants were individuals with knee OA (control and treatment) and healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Mild and moderate bilateral knee osteoarthritis
* Age between 50 and 70 years

Exclusion Criteria:

* Recent Lower limb injury
* Diabetic
* Knee or hip replacement
* Knees HA injection in last 6 months
* Any neuromuscular disease such as stroke and Parkinson

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Postural stability after treatment | baseline and 6 weeks
Changes in Biomechanics of gait after treatment | baseline and 6 weeks
Changes in biomechanics of stair climbing after treatment | baseline and 6 weeks

SECONDARY OUTCOMES:
Change in Pain after treatment | baseline and 6 weeks
Changes in WOMAC scores after treatment | baseline and 6 weeks

REFERENCES:
- [Derived] Khalaj N, Abu Osman NA, Mokhtar AH, George J, Abas WA. Effect of intra-articular hyaluronic injection on postural stability and risk of fall in patients with bilateral knee osteoarthritis. ScientificWorldJournal. 2014;2014:815184. doi: 10.1155/2014/815184. Epub 2014 Jun 19. PMID 25136689